CLINICAL TRIAL: NCT00745589
Title: Use of Sevelamer Hydrochloride to Control Hyperphosphatemia and Reduce Calcification Burden in the Poor Peritoneal Dialysis Patients
Brief Title: Sevelamer Hydrochloride in Peritoneal Dialysis Patients
Acronym: SERENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Dr., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A111-104
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Endstage Renal Disease
Keywords: vascular,; valvular calcification,; phosphate binder,; sevelamer,; endstage renal disease; peritoneal dialysis
MeSH Terms: interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- higher dose sevelamer (Active Comparator): first-line higher dose sevelamer hydrochloride
  Interventions: Drug: sevelamer hydrochloride
- low dose sevelamer (Active Comparator): second-line fixed low-dose sevelamer hydrochloride added to calcium carbonate
  Interventions: Drug: sevelamer hydrochloride

INTERVENTIONS:
Drug: sevelamer hydrochloride — First-line higher dose (that is, 800mg TDS and up to a maximum of 1200mg TDS) sevelamer hydrochloride will be compared against low dose second-line sevelamer hydrochloride (that is, fixed dose of 400mg TDS)
  Other Names: Renagel

SUMMARY:
To test the hypothesis that second-line fixed low-dose sevelamer hydrochloride therapy is as effective as first-line high-dose sevelamer hydrochloride therapy in limiting the progression of cardiovascular calcification.

DETAILED DESCRIPTION:
Cardiovascular disease accounts for nearly 50% of the mortality and is the most frequent cause of hospitalization in ESRD patients. Hyperphosphatemia is increasingly recognized to be an important predictor of mortality and cardiovascular death in ESRD patients and is largely attributed to the increased prevalence of vascular calcification.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients receiving long-term peritoneal dialysis treatment with hyperphosphatemia currently receiving aluminum-based phosphorus binders or whose phosphorus control remains suboptimal with calcium-based binders only
* Patients who cannot afford to self-pay sevelamer hydrochloride.
* Patients who provided informed consent for the study

Exclusion Criteria:

* Patients with underlying active malignancy
* Patients with cyanotic congenital heart disease
* Patients with poor general condition
* Patients with plan for living related kidney transplant within coming 1 year
* Female patients with pregnancy

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes in coronary artery, aortic valve, mitral annulus calcium scores | over 24 months
  Vascular and valvular calcium scores

SECONDARY OUTCOMES:
Changes in aortic pulse wave velocity | over 24 months
  arterial stiffness parameter
annualized percentage change in Coronary artery calcium score | over 12 months
  annualized percentage change in calcium score
Changess in serum T50 | over 24 months
  serum calcification propensity measure
Changes in serum calcium, phosphate | over 24 months
  biochemical parameters
Changes in alkaline phosphatase | over 24 months
  biochemical parameters
Changes in intact parathyroid hormone | over 24 months
  biochemical parameters
Changes in low density lipoprotein-cholesterol | over 24 months
  biochemical parameters
Changes in C-reactive protein | over 24 months
  biochemical parameters
Changes in systolic blood pressure | over 24 months
  blood pressure
Changes in diastolic blood pressure | over 24 months
  blood pressure
Changes in Forearm, femur and spine bone mineral density, T score and Z score | over 24 months
  Bone mineral density related parameters

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD, PhD, Principal Investigator — Queen Mary Hospital, University of Hong Kong
Locations (1):
- Queen Mary Hospital, Tung Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Wang AY, Pasch A, Wong CK, Chu IM, Tang TK, Chu J, Cheuk-Ying Fong C, Yau YY, Lo WK. Long-Term Effects of Sevelamer on Vascular Calcification, Arterial Stiffness, and Calcification Propensity in Patients Receiving Peritoneal Dialysis: The Randomized Pilot SERENE (Sevelamer on Vascular Calcification, Arterial Stiffness) Trial. Kidney Med. 2021 Nov 2;4(2):100384. doi: 10.1016/j.xkme.2021.10.002. eCollection 2022 Feb. PMID 35243302